CLINICAL TRIAL: NCT07239388
Title: Effectiveness of Structured Group Therapy in Reducing Depression and Anxiety Symptoms in Pakistan: A Randomised Controlled Trial
Brief Title: Structured Group Therapy in Reducing Depression and Anxiety in Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT_D_A_GT_2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adults; Anxiety
Keywords: Depression; Anxiety; Group therapy; Social support
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured group therapy (Experimental): This group will receive Cognitive Behavioural Therapy (CBT) and Mindfulness-Based Stress Reduction (MBSR) therapy techniques in group settings. The intervention will cover contents like: (1) Introduction to Depression and Anxiety: Understanding symptoms and causes; (2) Cognitive Restructuring: Identifying and challenging negative thoughts; (3) Stress Management: Techniques for managing physiological and psychological stress; (4) Mindfulness Practices: Meditation, breathing exercises, and body scanning; (5) Behavioural Activation: Planning and engaging in pleasurable and meaningful activities; (6) Social Support: Building and enhancing relationships; (7) Relapse Prevention: Strategies for maintaining progress after the intervention.
  Each group will consist of 8-10 participants to allow for optimal interaction and support. Twelve weekly group sessions, each lasting 90 minutes, will be conducted.
  Interventions: Other: Structured group therapy
- Treatment as usual (No Intervention): Participants will receive standard treatment or usual care, which may include individual therapy or medication, depending on their current treatment regimen.

INTERVENTIONS:
Other: Structured group therapy — Participants will receive Cognitive Behavioural Therapy (CBT) and Mindfulness-Based Stress Reduction (MBSR) therapy techniques in group settings. The intervention will cover contents like: (1) Introduction to Depression and Anxiety: Understanding symptoms and causes; (2) Cognitive Restructuring: Identifying and challenging negative thoughts; (3) Stress Management: Techniques for managing physiological and psychological stress; (4) Mindfulness Practices: Meditation, breathing exercises, and body scanning; (5) Behavioural Activation: Planning and engaging in pleasurable and meaningful activities; (6) Social Support: Building and enhancing relationships; (7) Relapse Prevention: Strategies for maintaining progress after the intervention.
  Each group will consist of 8-10 participants to allow for optimal interaction and support. Twelve weekly group sessions, each lasting 90 minutes, will be conducted.
  Arms: Structured group therapy

SUMMARY:
This study aims to assess the effectiveness of Cognitive Behavioural Therapy (CBT) and Mindfulness-Based Stress Reduction (MBSR) in group settings to reduce symptoms of depression and anxiety, enhance emotional resilience, and improve social support among Pakistani individuals struggling with these conditions.

DETAILED DESCRIPTION:
Mental health disorders, particularly depression and anxiety, are prevalent in Pakistan and significantly affect the emotional, social, and occupational well-being of individuals. According to the World Health Organisation (WHO), depression is the leading cause of disability globally, and anxiety disorders are among the most common mental health conditions in Pakistan, affecting millions.

In the Pakistani context, stigma surrounding mental illness, lack of awareness, and limited access to mental health services create substantial barriers to care. Group therapy, which provides a collective support system and skill-building strategies, can be an effective modality in addressing these challenges. Structured group therapy offers participants a sense of community, reduces feelings of isolation, and provides a platform for learning coping strategies within a culturally sensitive framework.

This study aims to assess the effectiveness of Cognitive Behavioural Therapy (CBT) and Mindfulness-Based Stress Reduction (MBSR) in group settings to reduce symptoms of depression and anxiety, enhance emotional resilience, and improve social support among Pakistani individuals struggling with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years)
* Diagnosed with moderate to severe depression
* Residing in urban or rural areas of Pakistan
* Willingness to attend 12 weekly group therapy sessions and comply with the study protocol

Exclusion Criteria:

* Severe psychiatric disorders (e.g., psychosis, bipolar disorder)
* Ongoing substance abuse or severe substance use disorder
* Participation in other therapeutic interventions (e.g., individual therapy or group therapy) during the study period
* Cognitive impairments that would interfere with participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Depression and anxiety | 12 weeks
  As measured through the participants' scores on the Hospital Anxiety & Depression Scale (HADS)

SECONDARY OUTCOMES:
Social support | 12 weeks
  As measured through participants' scores on the Multidimensional Scale of Perceived Social Support (MSPSS)
Functionality of participants | 12 weeks
  As measured through participants' scores on the WHO Disability Assessment Schedule (WHODAS 2.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No